CLINICAL TRIAL: NCT03432871
Title: The Role of Nicotinamide Riboside in Mitochondrial Biogenesis
Brief Title: Nicotinamide Riboside and Mitochondrial Biogenesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); Medical Research Council Mitochondrial Biology Unit (Unknown)
Responsible Party: Principal Investigator, Patrick Chinnery, Professor, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A094351
Record Dates: First submitted 2018-01-23; First posted 2018-02-14 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Mitochondrial Diseases; Mitochondrial Myopathies; Progressive External Ophthalmoplegia; Progressive Ophthalmoplegia; Progressive; Ophthalmoplegia, External; Mitochondria DNA Deletion; MELAS
Keywords: Mitochondria; Mitochondrial disease; Nicotinamide Riboside; Niagen; PEO; Single deletion; mtDNA deletion; MELAS; m.3243A>G
MeSH Terms: conditions — Mitochondrial Diseases; Mitochondrial Myopathies; Ophthalmoplegia, Chronic Progressive External; MELAS Syndrome | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Experimental medicine study (open label)
Masking Description: Experimental medicine study (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nicotinamide Riboside (Experimental): This is an open-label experimental medicine study.
  All subjects will receive the same dosage of the supplement Nicotinamide Riboside.
  Interventions: Dietary Supplement: Nicotinamide Riboside

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Nicotinamide Riboside is a member of the Vitamin B family which acts as a precursor to NAD+, an enzyme involved in energy production.
  Other Names: Niagen; Nicotinamide Riboside Chloride

SUMMARY:
Mitochondria are important parts of the cell that are responsible for producing energy. The amount of energy they produce depends on how much energy the body needs to function and this energy production can be severely impaired in people with mitochondrial disease. Symptoms of mitochondrial disease vary widely but usually involve the brain, nerves and muscles, as these are tissues that need a lot of energy. Mitochondrial disorders affect 1 in 5000 of the UK population and there is currently no cure.

Some scientists think that increasing the number of mitochondria in the body (mitochondrial biogenesis) might be an effective treatment for the symptoms of mitochondrial disease. Studies carried out in mice have shown that a type of B-vitamin called Nicotinamide Riboside (NR) is able to increase the number of mitochondria, leading to increased energy and a reduction in the symptoms of mitochondrial disease.

The aim of this study is to investigate if the same B vitamin, Nicotinamide Riboside, can increase energy production and reduce symptoms in humans with mitochondrial disease.

The study will consist of two parts:

Part 1: Participants will be given a single oral dose of Nicotinamide Riboside and the levels of NR in their bloodstream will be measured at regular intervals. This will involve a single overnight stay and simple blood tests.

Part 2: This requires 6 separate visits from each participant. Each participant will undergo a series of standard tests including a muscle biopsy and an MRI scan, then they will take a course of Nicotinamide Riboside (twice daily for 4 weeks). After 4 weeks of treatment, the participants will undergo the same tests again to see if there have been any changes in response to the treatment.

DETAILED DESCRIPTION:
Mitochondria are the primary source of energy within the cell, in the form of adenosine triphosphate (ATP). Mitochondrial ATP production is tightly regulated according to the energy requirements of the cell, but little is known about the underlying control mechanisms. This is important for the understanding of the biology of cell energetics and also relevant for patients with rare mitochondrial diseases where it has been proposed that inducing mitochondrial proliferation (biogenesis) might be an effective treatment. However, before embarking on therapeutic studies, it is essential to develop our understanding of the homeostatic mechanisms. Patients with mitochondrial diseases show an enhanced capacity for mitochondrial proliferation, and therefore provide an ideal platform to study mitochondrial homeostasis in vivo in man. The aim of this study, therefore, is to investigate the homeostatic mechanisms in this group of individuals because we are most likely to see an effect in this context.

Nicotinamide riboside (NR), a NAD+ natural precursor, boosts the PGC1α-dependent mitochondrial biogenesis pathway, leading to increased transcription of genes of the oxidative phosphorylation and improved motor performance of myopathic mice. This study is an open-label experimental medicine study using NR with the primary aim of determining whether there is mechanistic link between mitochondrial biogenesis and physiological function in humans with a similar mitochondrial disease.

This project consists of two studies, carried out in series. Both will investigate patients with a clinical and genetic diagnosis of:

i. Progressive external ophthalmoplegia (PEO) plus exercise intolerance/fatigue, caused by a single deletion of mitochondrial DNA

or

ii. Mitochondrial disease caused by the m.3243A>G mutation in mitochondrial DNA

Study 1: a 24 hour study before the experimental intervention, to confirm bioavailability of NR at a dosage within the range of a published study.

Patients (n=5) will be invited to the CRF for an overnight stay. If applicable, a urinary pregnancy test will be carried out before any study procedures commence. A baseline blood sample will be taken before administration of the supplement. Oral NR will be administered at a dosage of 10mg/kg -, and blood samples will be drawn at 30 mins,1, 2, 6, 12 and 24 hours post administration. These samples will be used for measurement of NR/NAD+ levels in blood at the relevant time points and ensure these are at expected levels before proceeding to experimental intervention.

Study 2: a 4-week study to determine whether NR induces mitochondrial biogenesis and affects mitochondrial function in patients with mitochondrial disease.

Patients (n=10) will undergo measurements of mitochondrial biogenesis and physiological activities. Oral NR will be administered at a dosage of 10mg/kg b.i.d, (taken twice daily, after food) and patients will be asked to return weekly for standard observations and to provide a blood sample. After 4 weeks of NR administration, patients will return for a repeat measure of the mitochondrial biogenesis parameters and physiological activities

ELIGIBILITY:
Inclusion Criteria:

Clinical and genetic diagnosis of:

* Progressive external ophthalmoplegia (PEO), caused by a single deletion of mitochondrial DNA
* or
* Mitochondrial disease caused by the m.3243A>G or A>T mutation in mitochondrial DNA
* Age 18-70 years
* Women of child-bearing age only if they are not pregnant or breast feeding at the inclusion into the study and agree not to become pregnant during the study. Female participants will undergo a pregnancy test before study commencement.
* Signed informed patient consent

Exclusion Criteria:

* Clinically significant liver disease (e.g., cirrhosis or a history of hepatitis)
* Presence of significant other neurological disorders (such as multiple sclerosis, Parkinson's disease) or major co-morbidities (such as definite cognitive impairment, psychiatric disease, heart or lung failure, orthopaedic or rheumatological disorders)
* Females who are at risk of pregnancy (i.e., not using regular contraception), who are pregnant, lactating or planning pregnancy
* Females taking the combined oral contraceptive pill (as oestrogens can induce mitochondrial biogenesis and interfere with study results)
* For MRI - medical contraindication e.g., pacemaker, deep brain stimulator, aneurysm clip or significant claustrophobia
* For biopsy - varicose veins overlying biopsy site, clinically significant lower limb oedema, active lower limb infection, use of anticoagulants or antiplatelet agents that cannot be discontinued, known bleeding diathesis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Bioavailability | Pharmacokinetic measure - 0, 0.5, 1, 2, 6, 12 and 24 hours post-dose
  Change in baseline levels of Nicotinamide Riboside detectable in the bloodstream of participants after a standard oral dose of the supplement (at 0, 0.5, 1, 2, 6, 12 and 24 hours)
Safety - Incidence of treatment related adverse events | 24 hours
  Observation over 24 hours after Nicotinamide Riboside administration. Recording of any adverse events or reactions
Safety - change in blood analytes | 24 hours
  Change from baseline in safety blood analyte levels - CK, Creatinine, Alanine Transaminase, Aspartate Transaminase (Units U/L)
Safety - temperature | Change measures - 0, 1, 2, 3, 4, 6, 8, 24 hours post-dose
  Change from baseline in patient temperature (degrees celsius, measurement at 0, 0.5, 1, 2, 6, 12 and 24 hours)
Safety - blood pressure | Change measures - 0, 1, 2, 3, 4, 6, 8, 24 hours post-dose
  Change from baseline in patient blood pressure (mmHg, measurement at 0, 0.5, 1, 2, 6, 12 and 24 hours)
Safety - pulse | Change measures - 0, 1, 2, 3, 4, 6, 8, 24 hours post-dose
  Change from baseline in patient pulse (bpm, measurement at 0, 0.5, 1, 2, 6, 12 and 24 hours)
Mitochondrial biogenesis - Magnetic Resonance Imaging | 4 weeks
  Change in in vivo measurement of mitochondrial function at the start and end of the 4 weeks of NR treatment (31P-MRS measurement of mitochondrial function - Phosphocreatine replenishment after exercise)
Mitochondrial biogenesis - Respiratory Chain Enzyme Analysis | 4 weeks
  Change from baseline in mitochondrial function at the start and end of the 4 weeks of NR treatment (Respiratory chain enzyme analysis)
Mitochondrial biogenesis - mitochondrial DNA quantification | 4 weeks
  Change from baseline in the amount of mitochondrial DNA at the start and end of the 4 weeks of NR treatment (mtDNA quantification)

SECONDARY OUTCOMES:
Impact on mitochondrial disease symptoms - Dynamometric measure of muscle strength | 4 weeks
  Participants will be asked to complete the dynamometric measure of muscle strength test, using a hand held dynamometer, before and after treatment. Force measured in kg.
Impact on mitochondrial disease symptoms - 6-minute walk | 4 weeks
  Participants will be asked to complete the 6 minute walk test before and after treatment. The distance they can walk in 6 minutes will be measured in metres.
Impact on mitochondrial disease symptoms - Quality of life (SF36 - qualitative) | 4 weeks
  Participants will be asked to complete the SF36 (Short Form 36) Quality of life questionnaire before and after treatment. This is a standard health survey used routinely in clinical practice.
Impact on mitochondrial disease symptoms - Timed get-up-and-go. | 4 weeks
  Participants will be asked to complete the Timed up and go test before and after treatment. The time taken to get up from sitting to standing will be measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Chinnery, Prof., Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No